CLINICAL TRIAL: NCT03221608
Title: Clinical Study of the Impact of Hyperthermic Intraperitoneal Chemotherapy on Peritoneal Recurrence and Prognosis of Patients With Stage T4 Colorectal Cancer After Radical Surgery: A Multicentre Randomised Clinical Trial
Brief Title: Clinical Analysis of HIPEC for T4 Colorectal Cancer After Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Second Affiliated Hospital, Sun Yat-Sen University (Other); Zhujiang Hospital (Other); First Affiliated Hospital of Jinan University (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Tcm-integrated Cancer Center of Southern Medical University (Unknown); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Nanfang Hospital, Southern Medical University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Donglin Ren, MD, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: zs6yhmjHIPEC2017
Record Dates: First submitted 2017-07-17; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Cancer; HIPEC; Peritoneal Carcinomatosis; Lobaplatin
MeSH Terms: conditions — Colorectal Neoplasms; Peritoneal Neoplasms | interventions — Surgical Procedures, Operative; Hyperthermic Intraperitoneal Chemotherapy; lobaplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery alone(open/laparoscopic) (Active Comparator): The patients with colorectal cancer (T4N0-2M0) who have a high risk of developing colorectal Peritoneal Carcinomatosis (PC) undergo curative surgery(open/laparoscopic).
  Interventions: Procedure: Surgery without HIPEC
- surgery and HIPEC (Experimental): Standard surgical treatment and HIPEC with Lobaplatin.
  Interventions: Procedure: Surgery and HIPEC with Lobaplatin

INTERVENTIONS:
Procedure: Surgery and HIPEC with Lobaplatin — The combination of surgery and HIPEC with Lobaplatin are performed in patients with colorectal cancer (T4N0-2M0).
  Other Names: The combination of surgery and HIPEC with Lobaplatin
  Arms: surgery and HIPEC
Procedure: Surgery without HIPEC — The patients with colorectal cancer (T4N0-2M0) are undergone a curative resection by laparoscopy or open approach.
  Other Names: Standard surgical treatment by laparoscopy or open approach.
  Arms: surgery alone(open/laparoscopic)

SUMMARY:
This multicentric study aims to determine if hyperthermic intraperitoneal chemotherapy (HIPEC) will help to prevent the development of peritoneal carcinomatosis in addition to the standard adjuvant systemic treatment after surgery.

DETAILED DESCRIPTION:
Background:

Colorectal cancer (CRC) is the third most common malignancy worldwide, nearly 1.4 million new cases every year, for about 694000 deaths. Surgery is the primary treatment and results in a cure rate of approximately 50% of the patients. However, recurrence following surgery is a major problem, the second most common site of recurrence was peritoneum, which was as a result of the intraperitioneal free cancer cells (FCC) and microscopic cancer (MC). The remaining free cancers and microscopic cancer in abdominal cavity can not be killed completely because of the "peritoneal-plasma barrier" and "non-sufficient drug concentration in abdominal cavity by systemic venous chemotherapy". In recent years, hyperthermic intraperitioneal chemotherapy(HIPEC) has already been shown to be effective in improving the 5 year survival rate of colorectal cancer. However, lots of clinically studies for patients with colorectal cancer are advanced, it is not sure yet whether surgery combined with HIPEC is effective on decreasing the rate of peritoneal carcinomatosis in T4 stage colorectal cancer. The efficacy tend to be magnified when stage T4 patients account for less, confusing HIPEC for treatment of patients with advanced colorectal cancer. Therefore, the aim of this study is to investigate the clinical efficacy of HIPEC in T4 stage patients, ruling out the effects of different T stages on curative effect. The results of this study will hopefully provide the clinical basis for improving the prognosis of patients with advanced colorectal cancer.

Study design： This is a multicenter study in which 300 patients with T4 colorectal cancer will be randomized to surveillance alone (control group) or HIPEC (experimental group) after resection of the primary tumor, either by laparoscopy or open approach. Subsequently, all patients started mfolfox6 chemotherapy after operation in a month. Adverse reaction of chemotherapy during chemotherapy and post chemotherapy period will be recorded.

Study population:

The patients with colorectal cancer (T4N0-2M0) will undergo a curative resection by laparoscopy or open approach.

Intervention:

HIPEC equipment used in the perfusion fluid (Lobaplatin of 50mg completely dissolved in 3000ml saline solution) is headed to 43℃. Then, it is injected into the peritoneal cavity by flow velocity of 200-400ml/min for 60 minutes.

Outcomes:

Primary endpoint is incidence of endoperitoneal recurrence at 36 months. Secondary endpoints are disease-free survival, overall survival, incidence of peritoneal carcinomatosis at end of follow-up with or without concomitant liver/lung metastases, quality of life and morbidity rate.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-proven colorectal adenocarcinoma
2. Patients with colon cancer or intraperitoneal rectal cancer with clinical (by CT) T4 tumors, any N, M0
3. Signed informed consent
4. White blood cell count of at least 3000/mm3, platelet count of at least 100.000/mm3
5. No bleeding diathesis or coagulopathy
6. Patients without chemotherapy, radiation or other anti-cancer treatment before the clinical trial

Exclusion Criteria:

1. Liver and/or lung metastases
2. Pregnant women or likely to be pregnant
3. Severe hepatic and / or renal dysfunction
4. Impossibility of an adequate follow-up
5. Without history of cancer during last 5 years
6. Other concurrent chemotherapy
7. Severe or uncontrolled mental illness
8. Patients with epilepsy required to be treated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of endoperitoneal recurrence at 36 months | 36 months

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 3 years
Disease-free survival (DFS) | 5 years
Overall survival (OS) | 3 years
Overall survival (OS) | 5 years
Quality of life | 3 years
  To evaluate quality of life with EORTC QLQ-30 questionnaire
HIPEC toxicity rate | 1 month
HIPEC toxicity rate | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: MeiJin Huang, MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University